CLINICAL TRIAL: NCT01861626
Title: Bioequivalence Study of V0057 Versus a Reference Formulation After Single Administration in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pierre Fabre Dermatology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: V00057 CA 1 01; 2013-000988-80 (EudraCT Number)
Record Dates: First submitted 2013-05-15; First posted 2013-05-23 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Isotretinoin

ARMS (2):
- sequence 1 : Test drug - Reference (Other)
  Interventions: Drug: V0057 - A mg; Drug: Isotretinoin
- Sequence 2 : Reference - Test drug (Other)
  Interventions: Drug: V0057 - A mg; Drug: Isotretinoin

INTERVENTIONS:
Drug: V0057 - A mg — Single oral administration
Drug: Isotretinoin — Single oral administration

SUMMARY:
The purpose of this study is to evaluate the bioequivalence (comparison of the rate and extent of the active substance into the body following single administration of the drugs) between the test product V0057 and a reference product after two single oral administration separate by 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject aged 18 to 50 years (inclusive)

Exclusion Criteria:

* Presence of any significant medical finding or significant history that may impact the safety, the interpretation of the results and/or the participation of the subject in the study according to the opinion of the investigator
* Presence of any clinically significant abnormal finding at examination in the Investigator's opinion

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 18 time points up to 72h after administration
Time of Maximum Concentration (Tmax) | 18 time points up to 72h after administration
Area under curve (AUC0-72) | 18 time points up to 72h after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Erfurt, Germany